CLINICAL TRIAL: NCT04722250
Title: SMall Annuli Randomized To Evolut™ or SAPIEN™ Trial
Acronym: SMART
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MDT20023EVR012
Record Dates: First submitted 2021-01-20; First posted 2021-01-25 (Actual); Results first posted 2025-03-20 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Symptomatic Aortic Stenosis; Aortic Valve Stenosis; Aortic Valve Replacement
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Medtronic Self-Expanding TAV (Experimental): Subjects will be randomized on a 1:1 basis to receive TAVR with either a Medtronic SE TAV or an Edwards BE THV.
  Interventions: Device: Medtronic Evolut PRO, Evolut PRO+ or Evolut FX (where commercially available) TAV Systems
- Edwards Balloon-Expandable THV (Experimental): Subjects will be randomized on a 1:1 basis to receive TAVR with either a Medtronic SE TAV or an Edwards BE THV.
  Interventions: Device: Edwards SAPIEN 3 or SAPIEN 3 Ultra THV Systems

INTERVENTIONS:
Device: Medtronic Evolut PRO, Evolut PRO+ or Evolut FX (where commercially available) TAV Systems — TAVR treatment with Medtronic Evolut PRO, PRO+ System or Evolut FX System (where commercially available)
  Arms: Medtronic Self-Expanding TAV
Device: Edwards SAPIEN 3 or SAPIEN 3 Ultra THV Systems — TAVR treatment with Edwards SAPIEN 3 or SAPIEN 3 Ultra System
  Arms: Edwards Balloon-Expandable THV

SUMMARY:
The purpose of this trial is to generate clinical evidence on valve safety and performance of self-expanding (SE) versus balloon-expandable (BE) transcatheter aortic valve replacement (TAVR) in subjects with a small aortic annulus and symptomatic severe native aortic stenosis.

Additionally, a stress echocardiography sub-study will be conducted as part of the SMART Trial at select sites. The purpose of the sub-study is to evaluate performance of SE versus BE TAVR in subjects with a small aortic annulus and symptomatic severe native aortic stenosis after undergoing exercise stress echocardiographic testing.

DETAILED DESCRIPTION:
This is a prospective, multi-center, international, randomized controlled, post-market trial.

The primary objectives of the trial are to demonstrate clinical non-inferiority and hemodynamic superiority of the Evolut PRO/PRO+/FX System when compared to subjects treated with the SAPIEN 3/3 Ultra System at 12 months post-procedure.

Subjects will be randomized on a 1:1 basis to receive TAVR with either a Medtronic SE Transcatheter Aortic Valve (TAV) or an Edwards BE Transcatheter Heart Valve (THV). Data will be collected at pre- and post-procedure, at discharge, at 30 days, and once a year until the 5-year follow-up is completed.

Product Names:

* Medtronic Evolut PRO and Evolut PRO+ TAV Systems, Evolut FX System (Commercially available in the United States and may be used upon commercial availability in Canada.)
* Edwards SAPIEN 3 and SAPIEN 3 Ultra THV Systems

The exercise stress echocardiographic testing at select SMART Trial sites seeks to evaluate the performance of the prosthetic aortic valve during exercise. The stress echocardiogram assessment will be conducted as part of the 12-month visit for participating subjects.

ELIGIBILITY:
Inclusion Criteria:

* Heart Team agrees that the subject is deemed symptomatic and is a candidate for transcatheter aortic valve replacement (TAVR)
* Subject has a predicted risk of operative mortality < 15% as determined by the local Heart Team
* Subject has severe aortic stenosis as determined by transthoracic echocardiography (TTE) at rest
* Subject has a small aortic annulus as determined by Multi-detector computed tomography (MDCT)
* Subject's anatomy is appropriate for both Medtronic Evolut PRO/PRO+/FX TAV and Edwards SAPIEN 3/3 Ultra TAV
* Subject's anatomy is suitable for TAVR via transfemoral vessel access
* Subject and the treating physician agree that the subject will return for all required post-procedure follow-up visits

Exclusion Criteria:

* Estimated life expectancy of fewer than 2 years
* Multivessel coronary artery disease with a Syntax score >32 and/or unprotected left main coronary artery(Syntax score calculation is not required for patients with history of previous revascularization if repeat revascularization is not planned).
* Participating in another trial that may influence the outcome of this trial
* Need for an emergent procedure for any reason
* Contraindicated for treatment with the Evolut PRO/PRO+/FX and Edwards SAPIEN 3/3 Ultra TAV in accordance with the Instructions for Use
* Other medical, social, or psychological conditions that in the opinion of the Investigator precludes the subject from appropriate consent or adherence to the protocol required follow-up exams
* Pregnant, nursing, or planning to be pregnant
* Subject is less than the legal age of consent, legally incompetent, unable to provide his/her own informed consent, or otherwise vulnerable
* Subject has an active COVID-19 infection or relevant history of COVID-19
* Previous aortic valve replacement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1103 (Actual)
Dates: Start 2021-04-02 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2027-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Herrmann, MD, Principal Investigator — University of Pennsylvania, United States; Roxana Mehran, MD, Principal Investigator — Mount Sinai School of Medicine, United States; Didier Tchétché, MD, Principal Investigator — Clinique Pasteur Toulouse, France
Locations (92):
- United States (61):
  - Scripps Memorial Hospital, La Jolla, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Sutter Health, San Francisco, California
  - Los Robles Hospital and Medical Center, Thousand Oaks, California
  - University of Colorado, Aurora, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - WHC Washington MedStar, Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - HealthPark Medical Center, Fort Myers, Florida
  - University of Florida, Gainesville, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Emory Structural Heart Clinic and Emory University Midtown, Atlanta, Georgia
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - NorthShore Health Systems, Evanston, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Saint Vincent Heart Center of Indiana, Carmel, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - AscensionVia Christi St. Francis Hospital, Wichita, Kansas
  - Tufts Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Ascension St. John Hospital, Detroit, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - St. Cloud Hospital, Saint Cloud, Minnesota
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Morristown Medical Center, Morristown, New Jersey
  - Buffalo General Medical Center, Buffalo, New York
  - NYU Langone Medical Center, New York, New York
  - The Icahn School of Medicine at Mount Sinai, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Memorial Hospital, Chapel Hill, North Carolina
  - TriHealth / Bethesda North Hospital, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Hillcrest Medical Center, Tulsa, Oklahoma
  - UPMC Pinnacle Harrisburg, Harrisburg, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - York Hospital, York, Pennsylvania
  - TriStar Centennial Medical Center, Nashville, Tennessee
  - St. Thomas West Hospital, Nashville, Tennessee
  - Seton Heart Institute, Austin, Texas
  - Baylor Jack and Jane Hamilton Heart and Vascular Hospital, Dallas, Texas
  - Texas Health Presbyterian Hospital/Dallas, Dallas, Texas
  - Baylor Saint Luke's Hospital, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - University of Texas Health Sciences Center at Houston - Center for Advanced Heart Failure, Houston, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - Intermountain Medical Center, Murray, Utah
  - Saint George Regional Hospital, St. George, Utah
  - University of Virginia, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - J.W. Ruby Memorial Hospital/West Virginia University, Morgantown, West Virginia
- Canada (5):
  - Providence Health-St. Paul's Hospital, Vancouver, British Columbia
  - Victoria Heart Institute Foundation/Royal Jubilee Hospital, Victoria, British Columbia
  - Toronto General Hospital, Toronto, Ontario
  - St. Michaels Hospital/Unity Health Toronto, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
- Rigshospitalet, Copenhagen, Denmark
- Helsinki University Hospital, Helsinki, Finland
- France (3):
  - Centre Hospitalier Universitaire de Clermont-Ferrand, Clermont-Ferrand
  - CHU Bordeaux, Pessac
  - Clinique Pasteur, Toulouse
- Germany (8):
  - Hers-und Diabeteszentrum NRW - Ruhr -Universitati Bochum, Bad Oeynhausen
  - Deutsches Herzzentrum Berlin, Berlin
  - Kath. St.-Johannes-Gesellschaft Dortmund gGmbH - St. Johannes-Hospital Dortmund, Dortmund
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Schleswig-Holstein - Campus Kiel, Kiel
  - Helios Health Institute GmbH, Leipzig
  - Universitätsklinikum Schleswig-Holstein - Campus Lübeck, Lübeck
  - Deutsches Herzzentrum Munchen, München
- Israel (2):
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (3):
  - Policlinico Sant' Orsala - Malpighi, Bologna
  - Azienda Ospedaliero-Universitaria Pisana - Stabilimento di Cisanello, Pisa
  - AOU Integrata Verona, Verona
- Netherlands (3):
  - Catharina Ziekenhuis, Eindhoven
  - Maastricht Universitair Medisch Centrum (MUMC), Maastricht
  - HagaZiekenhuis - Locatie Leyweg, The Hague
- Centro Hospitalar de Lisboa Ocidental, E.P.E. Hospital de Santa Cruz, Carnaxide, Portugal
- Hospital Vall d'Hebron, Barcelona, Spain
- Inselspital - Universitätsspital Bern, Bern, Switzerland
- United Kingdom (2):
  - Royal Infirmary of Edinburgh, Edinburgh
  - The Leeds Teaching Hospitals NHS Trust - Leeds General Infirmary, Leeds

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tchetche D, Mehran R, Blackman DJ, Khalil RF, Mollmann H, Abdel-Wahab M, Ben Ali W, Mahoney PD, Ruge H, Bleiziffer S, Lin L, Szerlip M, Grubb KJ, Byku I, Guerrero M, Gillam LD, Petronio AS, Attizzani GF, Batchelor WB, Gada H, Rogers T, Rovin JD, Whisenant B, Benton S, Gardner B, Padang R, Althouse AD, Herrmann HC. Transcatheter Aortic Valve Implantation by Valve Type in Women With Small Annuli: Results From the SMART Randomized Clinical Trial. JAMA Cardiol. 2024 Dec 1;9(12):1106-1114. doi: 10.1001/jamacardio.2024.3241. PMID 39382856
- [Derived] Herrmann HC, Mehran R, Blackman DJ, Bailey S, Mollmann H, Abdel-Wahab M, Ben Ali W, Mahoney PD, Ruge H, Wood DA, Bleiziffer S, Ramlawi B, Gada H, Petronio AS, Resor CD, Merhi W, Garcia Del Blanco B, Attizzani GF, Batchelor WB, Gillam LD, Guerrero M, Rogers T, Rovin JD, Szerlip M, Whisenant B, Deeb GM, Grubb KJ, Padang R, Fan MT, Althouse AD, Tchetche D; SMART Trial Investigators. Self-Expanding or Balloon-Expandable TAVR in Patients with a Small Aortic Annulus. N Engl J Med. 2024 Jun 6;390(21):1959-1971. doi: 10.1056/NEJMoa2312573. Epub 2024 Apr 7. PMID 38587261
- [Derived] Herrmann HC, Abdel-Wahab M, Attizzani GF, Batchelor W, Bleiziffer S, Verdoliva S, Chang Y, Gada H, Gillam L, Guerrero M, Mahoney PD, Petronio AS, Rogers T, Rovin J, Szerlip M, Whisenant B, Mehran R, Tchetche D. Rationale and design of the SMall Annuli Randomized To Evolut or SAPIEN Trial (SMART Trial). Am Heart J. 2022 Jan;243:92-102. doi: 10.1016/j.ahj.2021.09.011. Epub 2021 Sep 26. PMID 34587510

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1103 subjects were enrolled (consented): 212 subjects were exited prior to screening,154 exited the study prior to randomization, 737* subjects were randomized.
  *Notes: One additional subject was inadvertently randomized but was withdrawn after screening disapproval.
  -716 subjects had an attempted procedure, these subjects are the As-Treated set and are analyzed according to their first attempted device. This includes both administrative and procedural crossovers as shown below.
Period: Overall Study
Arm/Group | Medtronic Self-Expanding TAV | Edwards Balloon-Expandable THV
Started (Intention to treat (ITT) set according to subject randomization) | 366 | 371
Exited Prior to Procedure | 10 | 11
ITT (Intention to Treat) Population After Exit Prior to Procedure | 356 | 360
Administrative Cross-overs (Administrative cross-over subjects are those with first attempted procedure is with the other treatment device that they were not randomized to. These subjects are analyzed with the other treatment device in the as-treated set.) | 2 | 1
Attempted With Randomized Device | 354 | 359
Procedural Cross-overs (Procedural cross-overs are subjects who were first attempted with one device (per randomization assignment) and implanted with the other device at the time of the index procedure. These subjects are analyzed with the other treatment device in the implanted set.) | 4 | 0
Completed (Implanted with randomized device) | 350 | 359
Not Completed | 16 | 12

BASELINE CHARACTERISTICS:
Population: As Treated set (all subjects with attempted TAVR procedure according to first device used)
Groups:
- Total: Total of all reporting groups
Arm/Group | Medtronic Self-Expanding TAV | Edwards Balloon-Expandable THV | Total
Number analyzed (Participants) | 355 | 361 | 716
Age, Continuous [Mean (Standard Deviation); unit: years] | 80.1 (6.3) | 80.3 (6.1) | 80.2 (6.2)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender Female | 312 | 309 | 621
  Gender Male | 43 | 52 | 95
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity and race are reported only by US sites (SEV TAV n=183; BE TAV n= 184; Total N=367) This is for as treated subjects.
  **Note**: There are 8 SEV subjects and 5 BEV Subjects from US Sites who did not report ethnicity, therefore the total number with ethnicity reported are 175 SEV and 179 BEV.
  Participants
    Ethnicity of US Only, Unknown number also includes outside of US.: Hispanic or Latino | 4 | 5 | 9
    Ethnicity of US Only, Unknown number also includes outside of US.: Not Hispanic or Latino | 171 | 174 | 345
    Ethnicity of US Only, Unknown number also includes outside of US.: Unknown or Not Reported | 180 | 182 | 362
Race (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity and race are reported only by US sites (SEV TAV n=183; BE TAV n= 184; Total N=367) For as treated subjects.
  **NOTE**: There are 10 SEV subjects and 5 BEV subjects from US Sites that did not report race, therefore the total subjects are 173 SEV and 179 BEV.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 1 | 1 | 2
    Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
    Black or African American | 7 | 12 | 19
    White | 161 | 165 | 326
    More than one race | 2 | 1 | 3
    Unknown or Not Reported | 182 | 182 | 364
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 183 | 184 | 367
  United Kingdom | 18 | 18 | 36
  Switzerland | 1 | 1 | 2
  Portugal | 4 | 3 | 7
  Spain | 7 | 8 | 15
  Canada | 34 | 41 | 75
  Netherlands | 4 | 3 | 7
  Finland | 2 | 2 | 4
  Denmark | 3 | 4 | 7
  Italy | 18 | 18 | 36
  Israel | 6 | 7 | 13
  France | 16 | 15 | 31
  Germany | 59 | 57 | 116
Body Surface Area [Mean (Standard Deviation); unit: m^2] | 1.8 (0.2) | 1.8 (0.2) | 1.8 (0.2)
STS Score [Mean (Standard Deviation); unit: Percent] — Measure Description: The Society of Thoracic Surgeons (STS) Score is a score that represents the risk of operative mortality, major morbidity, and complications for adult cardiac surgeries.
  A total STS Score, presented as a risk probability on a scale of 0-100%, is calculated based on patient characteristics. The STS Score is calculated before a patient undergoes the transcatheter aortic valve replacement (TAVR) index procedure in the study, and a higher STS Score means a patient is at higher risk for surgery.
  Percent | 3.3 (1.9) | 3.2 (1.7) | 3.3 (1.8)
STS Category [Count of Participants; unit: Participants] — Patients are grouped into the following categories based on their STS score:
  <3, [3,5), [5,8), ≥ 8
  Participants
    Count of Participants | 355 | 361 | 716
    <3 | 182 | 191 | 373
    [3,5) | 122 | 123 | 245
    [5,8) | 37 | 35 | 72
    ≥ 8 | 14 | 12 | 26
NYHA (Baseline) [Count of Participants; unit: Participants] — New York Heart Association (NYHA) Class I: No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation or shortness of breath. Class II:Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, shortness of breath or chest pain. Class III:Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, shortness of breath or chest pain. Class IV: Symptoms of heart failure at rest. Any physical activity causes further discomfort.
  Participants
    NYHA I | 4 | 6 | 10
    NYHA II | 197 | 211 | 408
    NYHA III | 150 | 144 | 294
    NYHA IV | 4 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Mortality, Disabling Stroke or Heart Failure Rehospitalization
Description: Percentage of participants with all-cause mortality, disabling stroke, or heart failure rehospitalization.
Time Frame: 12 months
Population: As Treated set (all subjects with attempted TAVR procedure according to first device used)
Measure: Number; unit: Percent of Participants (K-M Rate)
Arm/Group | Medtronic Self-Expanding TAV | Edwards Balloon-Expandable THV
Number analyzed (Participants) | 355 | 361
Percent of Participants (K-M Rate) | 9.7 | 10.6
Statistical Analysis 1: Comparison: Medtronic Self-Expanding TAV vs Edwards Balloon-Expandable THV; Test type: Non-Inferiority — The endpoint is designed to test whether the Medtronic SE TAV is non-inferior to Edwards BE TAV in the composite event rate of all-cause mortality, disabling stroke or heart failure rehospitalization at 12 months post-procedure with an absolute non-inferiority margin of 8.0%; p < 0.001, z-test on Kaplan-Meier percentages; Risk Difference (RD) = -1.0, 90% CI 2-sided [-4.7 to 2.8]

2. Primary Outcome: Bioprosthetic Valve Dysfunction (BVD)
Description: Percentage of participants with BVD as determined by echocardiography (hemodynamic structural valve dysfunction (aortic valve no longer works properly as measured by hemodynamic mean gradient ≥ 20mmHg), non-structural valve dysfunction (severe prosthesis-patient mismatch (valve is too small) and/or ≥ moderate total aortic regurgitation (backward flow of blood)), thrombosis (formation of a blood clot), endocarditis (inflammation of the endocardium - the inner lining of the heart chambers and valves), or aortic valve re-intervention (a follow-up procedure to fix or replace the aortic prosthetic valve))
Time Frame: 12 months
Population: Implanted set (all subjects implanted with TAVR during index procedure according to last device implanted). *Note that a subject who is first attempted with one device then subsequently implanted with the other device will be analyzed according to the last implanted device.
Measure: Number; unit: Percent of Participants (K-M Rate)
Arm/Group | Medtronic Self-Expanding TAV | Edwards Balloon-Expandable THV
Number analyzed (Participants) | 350 | 365
Percent of Participants (K-M Rate) | 9.4 | 42.3
Statistical Analysis 1: Comparison: Medtronic Self-Expanding TAV vs Edwards Balloon-Expandable THV; Test type: Superiority; p < 0.001, z-test on Kaplan-Meier percentages; Risk Difference (RD) = -32.9, 95% CI 2-sided [-39.4 to -26.3]

3. Secondary Outcome: Percentage of Participants With BVD in Female Subjects
Description: as for outcome 2
Time Frame: 12 months
Population: Implanted set (all subjects implanted with TAVR during index procedure according to last device implanted) *Note that a subject who is first attempted with one device then subsequently implanted with the other device will be analyzed according to the last implanted device.
Measure: Number; unit: percentage of participants (K-M rate)
Arm/Group | Medtronic Self-Expanding TAV | Edwards Balloon-Expandable THV
Number analyzed (Participants) | 307 | 313
percentage of participants (K-M rate) | 8.4 | 42.7

4. Secondary Outcome: Percentage of Participants With Hemodynamic Structural Valve Dysfunction (HSVD)
Description: HSVD is defined as hemodynamic mean gradient ≥ 20mmHg on any echocardiogram after implant procedure.
Time Frame: 12 months
Population: as for outcome 3
Measure: Number; unit: percentage of participants (K-M rate)
Arm/Group | Medtronic Self-Expanding TAV | Edwards Balloon-Expandable THV
Number analyzed (Participants) | 350 | 365
percentage of participants (K-M rate) | 3.2 | 33.0

5. Secondary Outcome: Hemodynamic Mean Gradient as Continuous Variable
Description: Mean aortic gradient as measured by echocardiogram at the 12-month visit.
Time Frame: 12 months
Population: Implanted set (all subjects implanted with TAVR during index procedure according to last device implanted)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Medtronic Self-Expanding TAV | Edwards Balloon-Expandable THV
Number analyzed (Participants) | 298 | 301
mmHg | 7.7 (4.0) | 15.7 (6.7)

6. Secondary Outcome: Effective Orifice Area (EOA) as a Continuous Variable
Description: Effective Orifice Area (EOA) as measured by echocardiogram at the 12-month visit.
Time Frame: 12 months
Population: Implanted set (all subjects implanted with TAVR during index procedure according to last device implanted)
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | Medtronic Self-Expanding TAV | Edwards Balloon-Expandable THV
Number analyzed (Participants) | 267 | 266
cm2 | 1.98 (0.47) | 1.50 (0.35)

7. Secondary Outcome: Rate of Moderate or Severe Prothesis-patient Mismatch (PPM)
Description: Moderate or severe PPM will be defined as follows:
  For subjects with BMI < 30 kg/m2
  * Moderate PPM: EOAI = 0.85 - 0.65 cm2/m2
  * Severe PPM: EOAI = ≤ 0.65 cm2/m2
  For subjects with BMI ≥ 30 kg/m2
  * Moderate PPM: EOAI = 0.70 - 0.55 cm2/m2
  * Severe PPM: EOAI = ≤ 0.55 cm2/m2
Time Frame: 30 days
Population: Implanted set (all subjects implanted with TAVR during index procedure according to last device implanted)
Measure: Count of Participants; unit: Participants
Arm/Group | Medtronic Self-Expanding TAV | Edwards Balloon-Expandable THV
Number analyzed (Participants) | 273 | 296
Participants | 28 | 104

8. Other Pre Specified Outcome: Device Success
Description: Device Success is defined as meeting all of the following:
  Freedom from mortality AND Correct positioning of a single prosthetic heart valve into the proper anatomical location AND Intended performance of the prosthetic heart valve (no prosthesis-patient mismatch (PPM) and mean aortic valve gradient <20 mmHg or peak velocity <3 m/s) AND No moderate or severe prosthetic valve regurgitation)
Time Frame: 30 days
Population: As Treated set (all subjects with attempted TAVR procedure according to first device used)
Measure: Count of Participants; unit: Participants
Arm/Group | Medtronic Self-Expanding TAV | Edwards Balloon-Expandable THV
Number analyzed (Participants) | 291 | 319
Participants | 248 | 189

9. Other Pre Specified Outcome: Incidence of an Early Safety Composite
Description: Incidence of an early safety composite at 30 days defined as:
  * All-cause mortality
  * All stroke (disabling and non-disabling)
  * Life-threatening bleeding
  * Acute kidney injury-Stage 2 or 3 (including renal replacement therapy)
  * Coronary artery obstruction requiring intervention
  * Major vascular complication
  * Valve-related dysfunction requiring repeat procedure (BAV, TAVR, or SAVR)
Time Frame: 30 days
Population: As Treated set (all subjects with attempted TAVR procedure according to first device used)
Measure: Number; unit: percentage of participants (K-M rate)
Arm/Group | Medtronic Self-Expanding TAV | Edwards Balloon-Expandable THV
Number analyzed (Participants) | 355 | 361
percentage of participants (K-M rate) | 9.9 | 7.2

10. Other Pre Specified Outcome: Hospital Readmission Rate for Any Cause
Time Frame: 30 days
Population: As Treated set (all subjects with attempted TAVR procedure according to first device used)
Measure: Number; unit: percentage of participants (K-M rate)
Arm/Group | Medtronic Self-Expanding TAV | Edwards Balloon-Expandable THV
Number analyzed (Participants) | 355 | 361
percentage of participants (K-M rate) | 8.6 | 11.2

11. Other Pre Specified Outcome: Incidence of Clinical Efficacy
Description: Incidence of clinical efficacy (after 30 days) at 12 months defined as a composite of:
  * All-cause mortality
  * All stroke (disabling and non-disabling)
  * Requiring hospitalizations for valve-related symptoms or worsening congestive heart failure
  * NYHA class III or IV
  * Valve-related dysfunction (mean aortic valve gradient ≥20 mmHg, EOA ≤0.9-1.1 cm2 and/or Doppler velocity index (DVI) <0. 35m/s, AND/OR moderate or severe prosthetic valve regurgitation)
Time Frame: 12 months
Population: Implanted set (all subjects implanted with TAVR during index procedure according to last device implanted)
Measure: Number; unit: percentage of participants (K-M rate)
Arm/Group | Medtronic Self-Expanding TAV | Edwards Balloon-Expandable THV
Number analyzed (Participants) | 288 | 224
percentage of participants (K-M rate) | 12.5 | 31.5

12. Other Pre Specified Outcome: Percentage of Participants With Individual Clinical Endpoint Components Including Mortality, Disabling Stroke and Heart Failure Rehospitalization
Time Frame: 12 months and 2 Years
Population: As Treated set (all subjects with attempted TAVR procedure according to first device used)
Measure: Number; unit: percentage of participants (K-M rate)
Arm/Group | Medtronic Self-Expanding TAV | Edwards Balloon-Expandable THV
Number analyzed (Participants) | 355 | 361
percentage of participants (K-M rate)
  All Cause Mortality: 12 Months | 5.1 | 5.9
  Disabling Stroke: 12 Months | 3.1 | 2.6
  Heart Failure Rehospitalization: 12 Months | 4.1 | 3.5
  All Cause Mortality: 2 Years | 12.7 | 11.4
  Disabling Stroke: 2 Years | 4.7 | 3.2
  Heart Failure Rehospitalization: 2 Years | 6.1 | 6.0

13. Other Pre Specified Outcome: New Pacemaker Implantation Rate
Description: Note: This section is excluding subjects with pacemaker or ICD at baseline.
Time Frame: 30 days, 12 Months, 2 Years
Population: As Treated set (all subjects with attempted TAVR procedure according to first device used)
Measure: Number; unit: percentage of participants (K-M rate)
Arm/Group | Medtronic Self-Expanding TAV | Edwards Balloon-Expandable THV
Number analyzed (Participants) | 325 | 336
percentage of participants (K-M rate)
  30 Days | 12.1 | 7.8
  12 Months | 14.0 | 9.3
  2 Years | 15.4 | 11.4

14. Other Pre Specified Outcome: Aortic Valve Re-intervention Rate
Description: Aortic valve re-intervention rate as measured as the percentage of patients that had a procedure to fix or replace their prosthetic valve at the 30 days, 12 months and 2 Year visit.
Time Frame: 30 days, 12 months, 2 Years
Population: As Treated set (all subjects with attempted TAVR procedure according to first device used)
Measure: Number; unit: percentage of participants (K-M rate)
Arm/Group | Medtronic Self-Expanding TAV | Edwards Balloon-Expandable THV
Number analyzed (Participants) | 355 | 361
percentage of participants (K-M rate)
  30 Days | 0.6 | 0.3
  12 Months | 0.9 | 0.6
  2 Years | 0.9 | 0.9

15. Other Pre Specified Outcome: 6-minute Walk Test (6MWT) Change From Baseline
Time Frame: 30 days, 12 Months and 2 Years
Population: As Treated set (all subjects with attempted TAVR procedure according to first device used)
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Medtronic Self-Expanding TAV | Edwards Balloon-Expandable THV
Number analyzed (Participants) | 355 | 361
Meters
  30 Days | 25.5 (97.3) | 38.1 (86.7)
  12 Months | 39.5 (100.5) | 33.8 (94.8)
  2 Years | 29.5 (100.2) | 37.0 (90.1)

16. Other Pre Specified Outcome: Quality of Life (QoL) Change From Baseline (EuroQol- 5 Dimension [EQ-5D])
Description: EuroQol Group developed this Quality of Life (QOL) questionnaire referred to as EQ-5D that includes a descriptive system comprising five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
  The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. The answers given to ED-5D can be converted into EQ-5D index and utility scores anchored at 0 for death and 1 for perfect health. The EQ-5D Index Score is calculated for each study participant and the descriptive statistical summary of the EQ-5D score for the study population is provided. The EQ-5D Visual Analog Scale (VAS) Score is a scale numbered 0 to 100 (0 is the worse health the patient can imagine and 100 is the best health the patient can imagine).
Time Frame: 30 days, 12 Months and 2 Years
Population: As Treated set (all subjects with attempted TAVR procedure according to first device used)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medtronic Self-Expanding TAV | Edwards Balloon-Expandable THV
Number analyzed (Participants) | 355 | 361
score on a scale
  30 Days: EQ5D Index | 0.04 (0.15) | 0.05 (0.15)
  30 Days: EQ5D VAS | 8.1 (19.1) | 9.6 (19.7)
  12 Months: EQ5D Index | 0.04 (0.15) | 0.02 (0.15)
  12 Months: EQ5D VAS | 8.4 (20.1) | 7.6 (19.4)
  2 Years: EQ5D Index | 0.03 (0.15) | 0.02 (0.17)
  2 Years: EQ5D VAS | 8.2 (19.8) | 7.9 (19.6)

17. Other Pre Specified Outcome: Quality of Life (QoL) Change From Baseline (Kansas City Cardiomyopathy Questionnaire [KCCQ]
Description: Kansas City Cardiomyopathy Questionnaire (KCCQ): Quantifies physical function, symptoms, social function, selfefficacy and knowledge, and quality of life. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
  Note: This is the overall summary score for KCCQ.
Time Frame: 30 days, 12 Months and 2 Years
Population: As Treated set (all subjects with attempted TAVR procedure according to first device used)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medtronic Self-Expanding TAV | Edwards Balloon-Expandable THV
Number analyzed (Participants) | 355 | 361
score on a scale
  30 Days | 18.0 (19.4) | 17.7 (19.6)
  12 Months | 20.3 (20.3) | 17.6 (19.4)
  2 Years | 19.3 (20.1) | 17.3 (20.9)

18. Other Pre Specified Outcome: Bioprosthetic Valve Dysfunction (BVD)
Description: as for outcome 2
Time Frame: 2 Years
Population: Implanted set (all subjects implanted with TAVR during index procedure according to last device implanted).
Measure: Number; unit: percentage of participants (K-M rate)
Arm/Group | Medtronic Self-Expanding TAV | Edwards Balloon-Expandable THV
Number analyzed (Participants) | 350 | 365
percentage of participants (K-M rate) | 12.5 | 48.4

19. Other Pre Specified Outcome: Effective Orifice Area (EOA) as a Continuous Variable
Description: Effective Orifice Area (EOA) as measured by echocardiogram at the following intervals: Discharge, 30 Days, 12 Months and 2 Years
Time Frame: Discharge, 30 Days, 12 Months and 2 Years
Population: Implanted set (all subjects implanted with TAVR during index procedure according to last device implanted).
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Medtronic Self-Expanding TAV | Edwards Balloon-Expandable THV
Number analyzed (Participants) | 350 | 365
cm^2
  Discharge | 1.96 (0.43) | 1.63 (0.36)
  30 Days | 2.00 (0.46) | 1.52 (0.32)
  12 Months | 1.98 (0.47) | 1.50 (0.35)
  2 Years | 1.93 (0.48) | 1.51 (0.38)

20. Other Pre Specified Outcome: Hemodynamic Mean Gradient as a Continuous Variable
Description: Mean aortic gradient as measured by echocardiogram at the following intervals: Discharge, 30 Days, 12 Months and 2 Years
Time Frame: Discharge, 30 Days, 12 Months and 2 Years
Population: Implanted set (all subjects implanted with TAVR during index procedure according to last device implanted).
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Medtronic Self-Expanding TAV | Edwards Balloon-Expandable THV
Number analyzed (Participants) | 350 | 365
mmHg
  Discharge | 8.1 (3.7) | 14.8 (5.4)
  30 Days | 7.0 (3.1) | 14.4 (5.3)
  12 Months | 7.7 (4.0) | 15.7 (6.7)
  2 Years | 8.5 (4.2) | 16.1 (6.6)

21. Other Pre Specified Outcome: Rate of Paravalvular Leak (PVL) by Degree of Severity
Description: Paravalvular Leak as measured by the percentage of participants that had none, trace, mild, moderate and severe, at Discharge, 30 Days, 12 Months and 2 Years
Time Frame: Discharge, 30 Days, 12 Months and 2 Years
Population: Implanted set (all subjects implanted with TAVR during index procedure according to last device implanted).
Measure: Number; unit: percentage of participants
Arm/Group | Medtronic Self-Expanding TAV | Edwards Balloon-Expandable THV
Number analyzed (Participants) | 350 | 365
percentage of participants
  Discharge: PVL - None | 43.3 | 65.9
  Discharge: PVL - Trace | 43.9 | 28.9
  Discharge: PVL - Mild | 12.2 | 5.2
  Discharge: PVL - Moderate | 0.6 | 0.0
  Discharge: PVL - Severe | 0.0 | 0.0
  30 Days: PVL - None | 36.7 | 54.9
  30 Days: PVL - Trace | 46.0 | 32.5
  30 Days: PVL - Mild | 17.0 | 12.0
  30 Days: PVL - Moderate | 0.3 | 0.6
  30 Days: PVL - Severe | 0.0 | 0.0
  12 Months: PVL - None | 55.2 | 64.9
  12 Months: PVL - Trace | 30.6 | 15.5
  12 Months: PVL - Mild | 14.1 | 18.6
  12 Months: PVL - Moderate | 0.0 | 1.0
  12 Months: PVL - Severe | 0.0 | 0.0
  2 Years: PVL - None | 56.8 | 63.1
  2 Years: PVL - Trace | 27.6 | 18.8
  2 Years: PVL - Mild | 14.8 | 16.1
  2 Years: PVL - Moderate | 0.8 | 2.0
  2 Years: PVL - Severe | 0.0 | 0.0

22. Other Pre Specified Outcome: Mean Gradient ≥ 20 mmHg Based on Stress Echocardiogram
Description: Mean gradient ≥ 20 mmHg based on stress echocardiogram at select sites.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Medtronic Self-Expanding TAV | Edwards Balloon-Expandable THV
Number analyzed (Participants) | 29 | 33
Participants | 2 | 14

ADVERSE EVENTS:
Time Frame: Adverse Events were collected starting at the time the Informed Consent was signed through the primary endpoint snapshot. In this table we report all events from date of procedure through 2 Years post procedure for each subject.
Description: All serious adverse events S(AEs),non-serious endpoint-related AEs and adverse device effects (ADEs) that occurred during the study need to be reported throughout the trial duration. AEs are reported according to first device attempted at the TAVR procedure (As Treated Set). Subjects attempted with assigned device and subsequently implanted with the other device are also reported. *Note there were no non-serious events by MedDRA preferred term, that exceeded the 5% frequency threshold reporting
Groups:
- Attempted Medtronic Self-Expanding TAV (As Treated Set): Subjects will be randomized on a 1:1 basis to receive TAVR with either a Medtronic SE TAV or an Edwards BE THV.
  Medtronic Evolut PRO, Evolut PRO+ or Evolut FX (where commercially available) TAV Systems: TAVR treatment with Medtronic Evolut PRO, PRO+ System or Evolut FX System (where commercially available)
  **Note: As Treated set (all subjects with attempted TAVR procedure according to first device used)
- Attempted Edwards Balloon-Expandable THV (As Treated Set): Subjects will be randomized on a 1:1 basis to receive TAVR with either a Medtronic SE TAV or an Edwards BE THV.
  Edwards SAPIEN 3 or SAPIEN 3 Ultra THV Systems: TAVR treatment with Edwards SAPIEN 3 or SAPIEN 3 Ultra System
  **Note: As Treated set (all subjects with attempted TAVR procedure according to first device used)
- Attempted Both Devices: This arm contains subjects that had a procedural cross-over (i.e., subjects who were first attempted with one device (per randomization assignment) and implanted with the other device at the time of the index TAVR procedure).
  These subjects are analyzed with the other treatment device in the implanted set.
Arm/Group | Attempted Medtronic Self-Expanding TAV (As Treated Set) | Attempted Edwards Balloon-Expandable THV (As Treated Set) | Attempted Both Devices
All-Cause Mortality (participants affected / at risk) | 43/355 | 40/361 | 2/4
Serious Adverse Events (participants affected / at risk) | 210/355 | 207/361 | 4/4
Other Adverse Events (participants affected / at risk) | 0/355 | 0/361 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Attempted Medtronic Self-Expanding TAV (As Treated Set) (N=355) | Attempted Edwards Balloon-Expandable THV (As Treated Set) (N=361) | Attempted Both Devices (N=4)
Anaemia (Blood and lymphatic system disorders) | 12 (13) | 17 (19) | 1 (1)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (2) | 2 (2) | 0 (0)
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 5 (5) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0)
Acquired left ventricle outflow tract obstruction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 11 (11) | 8 (8) | 0 (0)
Angina pectoris (Cardiac disorders) | 3 (4) | 4 (4) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 2 (3) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 27 (28) | 29 (41) | 1 (1)
Atrial flutter (Cardiac disorders) | 4 (5) | 3 (3) | 0 (0)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block (Cardiac disorders) | 3 (3) | 3 (3) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 32 (34) | 17 (17) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 4 (4) | 1 (1) | 1 (1)
Bifascicular block (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0)
Bundle branch block left (Cardiac disorders) | 17 (17) | 15 (15) | 1 (1)
Bundle branch block right (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 3 (3) | 3 (3) | 0 (0)
Cardiac failure (Cardiac disorders) | 9 (12) | 15 (17) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 2 (2) | 4 (4) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 12 (16) | 10 (12) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 5 (5) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Cardiorenal syndrome (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Conduction disorder (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 2 (2) | 5 (6) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 4 (4) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Microvascular coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Mitral valve disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Mitral valve stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Nodal arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 5 (5) | 1 (1) | 0 (0)
Pericardial haemorrhage (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
Pulseless electrical activity (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 2 (2) | 5 (5) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Trifascicular block (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular dyssynchrony (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperparathyroidism primary (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Amaurosis fugax (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Angle closure glaucoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 1 (2) | 0 (0)
Corneal disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Macular degeneration (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Macular oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal artery occlusion (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (4) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Femoral hernia incarcerated (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric antral vascular ectasia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mesenteric arterial occlusion (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophageal achalasia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophageal food impaction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 2 (2) | 3 (3) | 0 (0)
Chest pain (General disorders) | 3 (3) | 3 (3) | 0 (0)
Death (General disorders) | 3 (3) | 6 (6) | 0 (0)
Device embolisation (General disorders) | 1 (1) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 2 (2) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperplasia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hypothermia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Impaired healing (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site extravasation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (3) | 5 (5) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
Prosthetic cardiac valve stenosis (General disorders) | 0 (0) | 2 (2) | 0 (0)
Prosthetic cardiac valve thrombosis (General disorders) | 2 (2) | 7 (7) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 0 (0)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Unevaluable event (General disorders) | 1 (1) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Amyloidosis (Immune system disorders) | 1 (1) | 1 (1) | 0 (0)
Sarcoidosis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Breast abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 5 (5) | 13 (14) | 0 (0)
Cellulitis (Infections and infestations) | 4 (4) | 1 (1) | 0 (0)
Clostridial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 2 (2) | 5 (6) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Enterococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Enterococcal sepsis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infective aneurysm (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Intervertebral discitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Metapneumovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 18 (20) | 16 (18) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Prosthetic valve endocarditis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Pseudomonal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyuria (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 7 (8) | 5 (5) | 0 (0)
Septic embolus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 4 (4) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Streptococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 8 (8) | 13 (13) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Vascular access site cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Vascular access site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Aortic pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 5 (6) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Incision site complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 (2) | 1 (1) | 0 (0)
Post procedural stroke (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Pseudomeningocele (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Shoulder fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) | 0 (0)
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vascular access site complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Vascular access site dissection (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Vascular access site haematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0)
Vascular access site occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vascular access site pseudoaneurysm (Injury, poisoning and procedural complications) | 5 (5) | 1 (1) | 0 (0)
Vascular access site rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Vascular procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Anticoagulation drug level above therapeutic (Investigations) | 1 (1) | 1 (1) | 0 (0)
Electrocardiogram P wave abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram PR prolongation (Investigations) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram QRS complex prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram ST segment elevation (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram change (Investigations) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Heart rate increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Myocardial necrosis marker increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Transvalvular pressure gradient increased (Investigations) | 0 (0) | 5 (5) | 0 (0)
Troponin increased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2) | 4 (4) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 (7) | 2 (2) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Vertebral column mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (4) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Hypergammaglobulinaemia benign monoclonal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebellar stroke (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 6 (6) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 14 (15) | 10 (10) | 2 (2)
Cervicogenic headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dementia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 3 (4) | 2 (2) | 0 (0)
Embolic stroke (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 3 (3) | 6 (6) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertensive encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0)
Reversible ischaemic neurological deficit (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal epidural haematoma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 4 (4) | 10 (10) | 0 (0)
Thalamic infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombotic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 3 (3) | 6 (8) | 0 (0)
Vascular dementia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 3 (6) | 0 (0) | 1 (1)
Device failure (Product Issues) | 2 (2) | 1 (1) | 0 (0)
Lead dislodgement (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Prosthetic cardiac valve failure (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Prosthetic cardiac valve malfunction (Product Issues) | 0 (0) | 8 (8) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 4 (4) | 0 (0)
Delirium (Psychiatric disorders) | 3 (3) | 2 (2) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Mental disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 3 (3) | 4 (7) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 11 (12) | 13 (16) | 0 (0)
Bladder mass (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (3) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal infarct (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urge incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 4 (4) | 0 (0) | 0 (0)
Breast haematoma (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 5 (5) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (4) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mediastinal haematoma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0)
Pleurocutaneous fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Peripheral artery bypass (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Aortic dissection (Vascular disorders) | 5 (5) | 0 (0) | 1 (1)
Arteriovenous fistula (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 4 (4) | 0 (0)
Femoral artery dissection (Vascular disorders) | 3 (3) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 8 (8) | 4 (4) | 0 (0)
Hypertensive crisis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Hypertensive emergency (Vascular disorders) | 1 (1) | 2 (2) | 0 (0)
Hypertensive urgency (Vascular disorders) | 2 (2) | 3 (4) | 0 (0)
Hypotension (Vascular disorders) | 5 (5) | 4 (4) | 0 (0)
Iliac artery dissection (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 2 (2) | 0 (0)
Pelvic venous thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 1 (2) | 1 (1) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Subclavian artery stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Subgaleal haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Superficial vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-12-15): https://cdn.clinicaltrials.gov/large-docs/50/NCT04722250/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-13): https://cdn.clinicaltrials.gov/large-docs/50/NCT04722250/SAP_001.pdf